CLINICAL TRIAL: NCT03954561
Title: Abdominal Compression Administered Early by the Colonoscopist Shortened Insertion Time of Water Exchange Colonoscopy
Brief Title: Abdominal Compression Administered Early by the Colonoscopist During Water Exchange Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Chief of Gastroenterology Endoscopy Suite, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: A10601001
Record Dates: First submitted 2017-06-10; First posted 2019-05-17 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Colonic Polyp; Colonic Adenoma
Keywords: colonoscopy; cecal intubation time
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopist group (Experimental): endoscopist-administered abdominal compression group
  Interventions: Procedure: endoscopist-administered abdominal compression
- assistant group (Active Comparator): assistant-administered abdominal compression group
  Interventions: Procedure: assistant-administered abdominal compression

INTERVENTIONS:
Procedure: endoscopist-administered abdominal compression — The endoscopist administers abdominal compression when loop formation encountered.
  Arms: endoscopist group
Procedure: assistant-administered abdominal compression — A assistant administers abdominal compression when loop formation encountered.
  Arms: assistant group

SUMMARY:
Loop formation is the most frequent cause of cecal intubation failure during colonoscopy. To reduce the loop formation, external abdominal pressure is widely used and proved to be helpful. Properly applied pressure can also decrease patients discomfort and shorten the cecal intubation time.

The loop formation during water exchange is less severe as compared with during air insufflation and can be reduced quite readily. Traditionally an assistant is not asked to administer abdominal compression until the endoscopist has struggled for some time and failed to reduce the loops by withdrawal. The colonoscopist can administer the abdominal compression whenever the scope is not advancing smoothly, probably in the early stage of loop formation. We test the hypothesis that colonoscopist administered abdominal compression to remove loops in their early stage of formation hastens cecal intubation.

A total of 120patients will be randomized in a 1:1 ratio (n=60 per group). When the tip of the scope doesn't advance or paradoxical movements occur, loop reduction by withdrawal of the scope will be implemented. If looping persists, abdominal compression will be applied. In the endoscopist-administered abdominal compression (endoscopist) group, the colonoscopist will apply the compression with his right hand and counter the pressure by pushing the back of the patient with his left forearm with the colonoscope in his left hand. The compression will be administered at left lower quadrant when the scope is in the sigmoid colon and at left lower quadrant and upper abdomen, respectively, when the scope tip reaches the transverse or ascending colon. If the formation of loop cannot be overcome, an assistant will apply the abdominal compression instead. In the assistant-administered abdominal compression (assistant) group, an endoscopic assistant will apply abdominal compression when a loop is formed. The assistant will apply the compression at the left lower quadrant initially, but quickly shift to other parts as needed depending on the tip location of colonoscope. If manual compressions fail, then the patients' position will be changed.

ELIGIBILITY:
Inclusion Criteria:

* In the Buddhist Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi, Taiwan.
* Patients who undergo WE colonoscopy performed by the two endoscopists (YHH and CWT) at the endoscopic suite will be included.

Exclusion Criteria:

* Included patient declined to give consent,
* age <20 years old,
* age >80 years old,
* previous partial colectomy, not completely consumed bowel prep regimen, massive ascites, or known colonic obstruction, morbid obesity (BMI ≥ 35).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
cecal intubation time | through study completion, average 15 minutes
  the time when the colonoscope is inserted from the anus to the cecum.

SECONDARY OUTCOMES:
proportion of patients requiring abdominal compression by an assistant | through study completion, average 15 minutes
  proportion of patients requiring abdominal compression by an assistant

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, MD, Principal Investigator — Buddhist Dalin Tzu Chi Hospital
Locations (1):
- Buddhist Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Rex DK, Goodwine BW. Method of colonoscopy in 42 consecutive patients presenting after prior incomplete colonoscopy. Am J Gastroenterol. 2002 May;97(5):1148-51. doi: 10.1111/j.1572-0241.2002.05681.x. PMID 12014719
- [Background] Shah SG, Brooker JC, Thapar C, Williams CB, Saunders BP. Patient pain during colonoscopy: an analysis using real-time magnetic endoscope imaging. Endoscopy. 2002 Jun;34(6):435-40. doi: 10.1055/s-2002-31995. PMID 12048623
- [Background] Herreros de Tejada A, Gimenez-Alvira L, Van den Brule E, Sanchez-Yuste R, Matallanos P, Blazquez E, Calleja JL, Abreu LE. Severe splenic rupture after colorectal endoscopic submucosal dissection. World J Gastroenterol. 2014 Jul 28;20(28):9618-20. doi: 10.3748/wjg.v20.i28.9618. PMID 25071360
- [Background] Waye JD, Yessayan SA, Lewis BS, Fabry TL. The technique of abdominal pressure in total colonoscopy. Gastrointest Endosc. 1991 Mar-Apr;37(2):147-51. doi: 10.1016/s0016-5107(91)70673-1. PMID 2032597
- [Background] Church JM. Ancillary colonoscope insertion techniques. An evaluation. Surg Endosc. 1993 May-Jun;7(3):191-3. doi: 10.1007/BF00594106. PMID 8503077
- [Background] Catalano F, Catanzaro R, Branciforte G, Bentivegna CF, Cipolla R, Brogna A, Sala LO, Migliore G, Paternuosto M. Colonoscopy technique with an external straightener. Gastrointest Endosc. 2000 May;51(5):600-4. doi: 10.1016/s0016-5107(00)70301-4. PMID 10805853
- [Background] Tsutsumi S, Fukushima H, Kuwano H. Colonoscopy using an abdominal bandage. Hepatogastroenterology. 2007 Oct-Nov;54(79):1983-4. PMID 18251143
- [Background] Dechene A, Jochum C, Bechmann LP, Windeck S, Gerken G, Canbay A, Zopf T. Magnetic endoscopic imaging saves abdominal compression and patient pain in routine colonoscopies. J Dig Dis. 2011 Oct;12(5):364-70. doi: 10.1111/j.1751-2980.2011.00524.x. PMID 21955429
- [Background] Hsieh YH, Tseng KC, Chou AL. Patient self-administered abdominal pressure to reduce loop formation during minimally sedated colonoscopy. Dig Dis Sci. 2010 May;55(5):1429-33. doi: 10.1007/s10620-009-0876-3. Epub 2009 Jul 7. PMID 19582577
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Hsieh YH, Koo M, Leung FW. A patient-blinded randomized, controlled trial comparing air insufflation, water immersion, and water exchange during minimally sedated colonoscopy. Am J Gastroenterol. 2014 Sep;109(9):1390-400. doi: 10.1038/ajg.2014.126. Epub 2014 Jun 3. PMID 24890443
- [Background] Cadoni S, Sanna S, Gallittu P, Argiolas M, Fanari V, Porcedda ML, Erriu M, Leung FW. A randomized, controlled trial comparing real-time insertion pain during colonoscopy confirmed water exchange to be superior to water immersion in enhancing patient comfort. Gastrointest Endosc. 2015 Mar;81(3):557-66. doi: 10.1016/j.gie.2014.07.029. Epub 2014 Sep 26. PMID 25262100
- [Background] Jia H, Pan Y, Guo X, Zhao L, Wang X, Zhang L, Dong T, Luo H, Ge Z, Liu J, Hao J, Yao P, Zhang Y, Ren H, Zhou W, Guo Y, Zhang W, Chen X, Sun D, Yang X, Kang X, Liu N, Liu Z, Leung F, Wu K, Fan D. Water Exchange Method Significantly Improves Adenoma Detection Rate: A Multicenter, Randomized Controlled Trial. Am J Gastroenterol. 2017 Apr;112(4):568-576. doi: 10.1038/ajg.2016.501. Epub 2016 Dec 6. PMID 27922025
- [Background] Hsieh YH, Tseng CW, Hu CT, Koo M, Leung FW. Prospective multicenter randomized controlled trial comparing adenoma detection rate in colonoscopy using water exchange, water immersion, and air insufflation. Gastrointest Endosc. 2017 Jul;86(1):192-201. doi: 10.1016/j.gie.2016.12.005. Epub 2016 Dec 15. PMID 27988288
- [Background] Rex DK. Water exchange vs. water immersion during colonoscope insertion. Am J Gastroenterol. 2014 Sep;109(9):1401-3. doi: 10.1038/ajg.2014.235. PMID 25196871
- [Background] Leung JW, Thai A, Yen A, Ward G, Abramyan O, Lee J, Smith B, Leung F. Magnetic endoscope imaging (ScopeGuide) elucidates the mechanism of action of the pain-alleviating impact of water exchange colonoscopy - attenuation of loop formation. J Interv Gastroenterol. 2012 Jul;2(3):142-146. doi: 10.4161/jig.23738. Epub 2012 Jul 1. PMID 23805397
- [Background] Kudo Se, Lambert R, Allen JI, Fujii H, Fujii T, Kashida H, Matsuda T, Mori M, Saito H, Shimoda T, Tanaka S, Watanabe H, Sung JJ, Feld AD, Inadomi JM, O'Brien MJ, Lieberman DA, Ransohoff DF, Soetikno RM, Triadafilopoulos G, Zauber A, Teixeira CR, Rey JF, Jaramillo E, Rubio CA, Van Gossum A, Jung M, Vieth M, Jass JR, Hurlstone PD. Nonpolypoid neoplastic lesions of the colorectal mucosa. Gastrointest Endosc. 2008 Oct;68(4 Suppl):S3-47. doi: 10.1016/j.gie.2008.07.052. No abstract available. PMID 18805238
- [Background] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102